CLINICAL TRIAL: NCT02561312
Title: Comparison of Two Methods of Transfusion for Stroke Prevention in Sickle Cell
Status: Completed | Type: Observational
Sponsor: Chattanooga-Hamilton County Hospital Authority (Other)
Responsible Party: Principal Investigator, Jennifer Keates, M.D., Pediatric Oncologist / Hematologist, Chattanooga-Hamilton County Hospital Authority
Other Study IDs: 15-084
Record Dates: First submitted 2015-09-23; First posted 2015-09-28 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Anemia, Sickle Cell; Sickling Disorder Due to Hemoglobin S
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RMPET: For rapid manual partial exchange transfusion, participants with a weight >50kg, 500 ml of whole blood is removed from the participant via a single lumen central venous line, followed by infusion of 500 ml of saline. A 30 second wait time is utilized for equilibration to occur. A second 500 ml aliquot is removed, and then two units of packed red blood cells (PRBC) are infused. (This is customized for a patient with large red blood cell mass). For participants <50 kg, the individual exchange aliquots are adjusted to 10 ml/kg or normal saline and PRBC.
  Interventions: Other: Rapid manual partial exchange transfusion
- Simple Transfusion: For simple transfusion, the volume of packed red blood cells (PRBC) to be transfused in the participant is 10-15 cc/kg. No normal saline exchange is required. All blood is transfused through a single lumen central venous line.
  Interventions: Other: Simple Transfusion

INTERVENTIONS:
Other: Rapid manual partial exchange transfusion — The first four participants will receive peripheral red blood cells via rapid manual partial exchange transfusions every month for 6 months. There is a pre-study washout for 3 months then there is a 3 month test period (data collection) before the participant is transferred to ST treatment.
  Groups: RMPET
Other: Simple Transfusion — The second group of four participants will receive peripheral red blood cells via simple transfusion every month for 6 months. There is a pre-study washout period for 3 months then there is a 3 month test period (data collection) before the participant is transferred to RMPET treatment.
  Groups: Simple Transfusion

SUMMARY:
Chronic blood transfusions are essential supportive care for sickle cell patients at high risk for morbidity and mortality due to stroke. These patients, however, are at risk for iron overload. In the investigator's comprehensive sickle cell center, the investigators support chronic transfusion with rapid manual partial exchange transfusions (RMPET) using a single access central line port. The investigators do not have a comprehensive adult sickle cell program but upon transition of patients the patients would be provided simple transfusion (ST) in an adult ambulatory infusion setting due to nursing acuity needed for RMPET. The investigators plan to study the institution's participants currently on chronic transfusion support and compare different transfusion modalities to better understand the effects from switching from RMPET to ST. To date, there are no such comparisons within and between sickle cell patients in the literature.

DETAILED DESCRIPTION:
II. Objective. Compare differences in RMPET versus ST.

III. Specific Aims:

1. To compare key predictive hematologic factors (hematocrit, hemoglobin, hemoglobin S quantification, blood volume and alloantibodies) for relative risk of stroke utilizing two methods of blood transfusion therapy.
2. To determine the nursing time to administer straight versus manual exchange transfusion therapy.
3. To survey patient satisfaction for both procedures.

IV: Background/Significance:

Stroke occurs in 10% of Sickle Cell Disease (SCD) patients before the age of 20 Years. Current standard of care for secondary overt stroke prevention in patients with SCD is chronic red blood cell (RBC) transfusions. Stroke recurs in ~ 60% of patients without chronic RBC therapy and in ~ 20% of patients with chronic transfusion while maintaining a hemoglobin S percentage of less than 30%. Indefinite transfusion therapy is practiced as discontinuation after short-term or long-term prophylactic transfusions leads to recurrent overt strokes and more ensuing CNS damage, even with transition to hydroxyurea. Chronic transfusions also prevent initial stroke in high-risk patients identified by transcranial Doppler (TCD) ultrasound. The Stroke Prevention Study in Sickle Cell Disease (STOP) demonstrated a 92% stroke risk reduction among 63 of 130 children with abnormal TCD results. Rates of stroke declined significantly since implementing routine TCD screening and primary prophylactic transfusion therapy. The subsequent STOP 2 trial supports the use of chronic transfusion indefinitely because discontinuation resulted in an increased rate of abnormal TCD conversion and development of overt stroke. Discontinuing transfusions on the STOP 2 trial was also associated with a higher occurrence of silent cerebral infarcts, documented in 3 of 37 patients (8.1%) in the continued-transfusion group compared with 11 of 40 (27.5%) in the transfusion-halted group. More recent studies demonstrate that SCD patients are also at risk for silent cerebral infarcts. An association between worsening vasculopathy shown by magnetic resonance angiography and progressive overt and silent infarcts on magnetic resonance imaging has been found. More aggressive magnetic resonance imaging screening may be indicated and this could result in more patients with SCD treated with chronic transfusion.

Common chronic transfusion modalities include ST or RMPET. The goal of therapy is to reduce the hemoglobin S level either by diluting the blood (ST) or by removing and replacing the blood with non-sickle hemoglobin (RMPET). To prevent further brain injury, the goal of transfusion therapy is to lower the hemoglobin S quantification to less than 30% on a routine basis, usually monthly transfusion procedure. There are many large centers that utilize erythrocytapheresis which is considered the preferable method if available.

The investigator's study will focus on the types of RBC exchange therapy currently utilized in the investigator's Infusion Clinic at T.C. Thompson Children's Hospital. The investigators will determine which transfusion method is best for each participant for achieving the hematologic parameters of lower hemoglobin S quantification.The investigators will also measure the amount of nursing time for each procedure and which method is preferred by participants. The investigators will share the institutional observations with other institutions who may intend to switch between RMPET and ST.

V. Methods:

Study Design: Prospective observational cohort study

The investigators will utilize the institution's current population of 8 eligible chronically exchanged transfused participants at the T.C. Thompson Children's Infusion Clinic. The eligible participants will be invited to participate in a cross over design study so that each participant serves as its own control. Eight participants will be randomly assigned (blinded envelope) whereby four participants will start with rapid manual partial exchange transfusion: 3 months will be spent in a wash out period, then 3 months of data collection for RMPET. This group will then be switched to simple transfusion with a wash out period of three months, then data collection for three months. The second group of four participants will start with simple transfusion and have an identical study design over 12 months (3 months of collected data during simple transfusion, a 3 month wash out period, switch to rapid manual partial exchange transfusion for three months, then 3 months of data collection for RMPET).

The investigators will optimize all therapy to achieve the post transfusion goal of <30% hemoglobin S and post transfusion Hb <12g/DL.with each transfusion performed for best practice in avoiding sickle cell complications.

ELIGIBILITY:
Inclusion Criteria:

1. Participants between 3 and 25 years of age
2. Diagnosis of Hemoglobin SS or SBeta thalassemia
3. On chronic exchange for stroke prevention
4. Performance status: Lansky play score of 100%, and if over 16 years of age, Karnofsky=100%

Exclusion Criteria:

1. Participant has experienced more than one stroke and has a modified Rankin Scale of >3.
2. Diagnosis of Hemoglobin SC disease
3. Participants on chronic transfusion for priapism.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 8 chronically exchanged transfused participants at T.C. Thompson Children's Infusion Clinic with sickle cell disease (Hemoglobin SS or SBeta thalassemia) currently receiving rapid manual partial exchange transfusion.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Hemoglobin S, baseline hemoglobin/hematocrit, | Pre Infusion, lab collected monthly for one year thru study completion
  Lab parameters pre-infusion for each method of transfusion

SECONDARY OUTCOMES:
Hemoglobin S, end of transfusion hemoglobin/hematocrit, blood volume, alloantibodies, | Post Infusion, lab collected monthly for one year thru study completion
  Lab parameters post-infusion for each method of transfusion

OTHER OUTCOMES:
Nursing Time score | Monthly at end of each transfusion for one year thru study completion
  Determine nursing time to administer straight versus manual exchange transfusion
Patient Satisfaction Questionnaire | At end of 6 month period and at 12 months (after RMPET and ST)
  Patient satisfaction questionnaire consisting of 5 Likert scaled questions for preference of RMPET versus ST assessed after six months on either cohort

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Keates, MD, Principal Investigator — Children's Hospital at Erlanger
Locations (1):
- Chidlren's Hospital at Erlanger, Chattanooga, Tennessee, United States

REFERENCES:
- [Background] Scothorn DJ, Price C, Schwartz D, Terrill C, Buchanan GR, Shurney W, Sarniak I, Fallon R, Chu JY, Pegelow CH, Wang W, Casella JF, Resar LS, Berman B, Adamkiewicz T, Hsu LL, Ohene-Frempong K, Smith-Whitley K, Mahoney D, Scott JP, Woods GM, Watanabe M, Debaun MR. Risk of recurrent stroke in children with sickle cell disease receiving blood transfusion therapy for at least five years after initial stroke. J Pediatr. 2002 Mar;140(3):348-54. doi: 10.1067/mpd.2002.122498. PMID 11953734
- [Background] Hulbert ML, McKinstry RC, Lacey JL, Moran CJ, Panepinto JA, Thompson AA, Sarnaik SA, Woods GM, Casella JF, Inusa B, Howard J, Kirkham FJ, Anie KA, Mullin JE, Ichord R, Noetzel M, Yan Y, Rodeghier M, Debaun MR. Silent cerebral infarcts occur despite regular blood transfusion therapy after first strokes in children with sickle cell disease. Blood. 2011 Jan 20;117(3):772-9. doi: 10.1182/blood-2010-01-261123. Epub 2010 Oct 12. PMID 20940417
- [Background] Ware RE, Helms RW; SWiTCH Investigators. Stroke With Transfusions Changing to Hydroxyurea (SWiTCH). Blood. 2012 Apr 26;119(17):3925-32. doi: 10.1182/blood-2011-11-392340. Epub 2012 Feb 7. PMID 22318199
- [Background] Adams RJ, McKie VC, Hsu L, Files B, Vichinsky E, Pegelow C, Abboud M, Gallagher D, Kutlar A, Nichols FT, Bonds DR, Brambilla D. Prevention of a first stroke by transfusions in children with sickle cell anemia and abnormal results on transcranial Doppler ultrasonography. N Engl J Med. 1998 Jul 2;339(1):5-11. doi: 10.1056/NEJM199807023390102. PMID 9647873
- [Background] Enninful-Eghan H, Moore RH, Ichord R, Smith-Whitley K, Kwiatkowski JL. Transcranial Doppler ultrasonography and prophylactic transfusion program is effective in preventing overt stroke in children with sickle cell disease. J Pediatr. 2010 Sep;157(3):479-84. doi: 10.1016/j.jpeds.2010.03.007. PMID 20434165
- [Background] McCarville MB, Goodin GS, Fortner G, Li CS, Smeltzer MP, Adams R, Wang W. Evaluation of a comprehensive transcranial doppler screening program for children with sickle cell anemia. Pediatr Blood Cancer. 2008 Apr;50(4):818-21. doi: 10.1002/pbc.21430. PMID 18085672
- [Background] McCavit TL, Xuan L, Zhang S, Flores G, Quinn CT. National trends in incidence rates of hospitalization for stroke in children with sickle cell disease. Pediatr Blood Cancer. 2013 May;60(5):823-7. doi: 10.1002/pbc.24392. Epub 2012 Nov 14. PMID 23151905
- [Background] Adams RJ, Brambilla D; Optimizing Primary Stroke Prevention in Sickle Cell Anemia (STOP 2) Trial Investigators. Discontinuing prophylactic transfusions used to prevent stroke in sickle cell disease. N Engl J Med. 2005 Dec 29;353(26):2769-78. doi: 10.1056/NEJMoa050460. PMID 16382063
- [Background] Casella JF, King AA, Barton B, White DA, Noetzel MJ, Ichord RN, Terrill C, Hirtz D, McKinstry RC, Strouse JJ, Howard TH, Coates TD, Minniti CP, Campbell AD, Vendt BA, Lehmann H, Debaun MR. Design of the silent cerebral infarct transfusion (SIT) trial. Pediatr Hematol Oncol. 2010 Mar;27(2):69-89. doi: 10.3109/08880010903360367. PMID 20201689